CLINICAL TRIAL: NCT05883943
Title: First-in-Human Early Feasibility Clinical Evaluation of Safety, Efficacy and Utility of the Cook® Venous Valve System for Treatment of Chronic Venous Insufficiency
Brief Title: Cook Venous Valve System for Treatment of Chronic Venous Insufficiency
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MED Institute Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-4344
Record Dates: First submitted 2023-05-15; First posted 2023-06-01 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Venous Insufficiency of Leg

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Cook® Venous Valve System (Experimental)
  Interventions: Device: Cook® Venous Valve System

INTERVENTIONS:
Device: Cook® Venous Valve System — The Cook® Venous Valve is a permanent prosthetic, bicuspid, one-way flow valve designed to be percutaneously implanted into the peripheral deep venous system. The Cook® Venous Valve Delivery System is used to percutaneously deliver the Cook® Venous Valve into the deep venous system.

SUMMARY:
The purpose of this study is to learn about the safety, efficacy and utility of a medical device called the Cook® Venous Valve System. This device, percutaneously placed in the leg, is meant to help the blood flow correctly through the veins in the leg.

ELIGIBILITY:
Limited inclusion criteria:

* Documented symptomatic deep venous reflux in one limb
* Deep venous reflux in the region of interest

Limited exclusion criteria:

General:

* Age < 18 years
* BMI ≥ 40
* Cultural objections to porcine materials
* Unwillingness or inability to comply with the follow-up
* Unwillingness to provide study data for duration of study
* Simultaneous participation in another device or drug study
* Inability or refusal to give informed consent

Medical:

* Pregnant, or planning to become pregnant
* Diagnosis of terminal illness with life expectancy less than 12 months
* Complete symptom resolution with compliant compression therapy for three months
* Untreated superficial venous disease
* Medical interventions including any of the following: planned procedure of any leg, vascular intervention or major surgery within the last three months, implanted inferior vena cava filter
* Medical history of any of the following: anticoagulation treatment for pulmonary embolism (within the last six months or ongoing), insulin dependent diabetes, chronic obstructive pulmonary disease, renal dysfunction requiring dialysis, leg amputation, bleeding diathesis, untreated or unresolved systemic infection or local infection, active malignancy except non-melanoma skin cancer, other acute or chronic medical condition that may cause noncompliance with the protocol or confound the study results, documented history of significant untreated stenosis within the arterial system
* Positive coronavirus (COVID-19) test six days prior to implant procedure

Anatomical:

* Inability to clearly visualize target implantation site
* Tortuous target implantation site
* Inadequate inflow and/or outflow to the target region

Procedural:

* Inability to gain access to the access site vein
* Untreated focal or diffuse stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2023-09-23 (Actual); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Freedom from major adverse events in the first 30 days | 30 days after enrollment
  The primary safety endpoint is freedom from major adverse events (MAE) in the first 30 days, where MAE is defined as: death, clinically-driven reintervention, bleeding requiring transfusion, flow limiting dissection of the target vessel, or clinically significant deep vein thrombosis (DVT), pulmonary embolism, or device migration.

SECONDARY OUTCOMES:
Freedom from MAE at three months, six months, and 12 months | Three months, six months, and 12 months after enrollment
  The secondary safety endpoint is freedom from MAE at three months, six months, and 12 months.

CONTACTS AND LOCATIONS:
Locations (3):
- Colombia (3):
  - Angiosur S.A.S., Antioquia
  - Clínica de La Costa S.A.S., Barranquilla
  - Fundacion Oftalmologica De Santander, Santander

IPD SHARING:
Plan to Share IPD: No